CLINICAL TRIAL: NCT02927041
Title: Observational Prospective Transesophageal Myocardial Ultrasound Survey
Acronym: OPTEMUS
Status: Withdrawn | Type: Observational
Why Stopped: Funding and supplies ran out
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Memorial Hermann Health System (Other)
Responsible Party: Principal Investigator, yafen liang, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-16-0376
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hemodynamic Instability
Keywords: hemodynamic transesophageal echocardiography
MeSH Terms: interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- OR-Trauma: Patients presenting with hemodynamic instability with expected intubation greater than 24 hours. Hemodynamic monitoring with transesophageal echo and hemodynamic support/ interventions include volume resuscitation, vasopressors, and positive inotropes. The Anesthesiologist may or may not use the information provided by the transesophageal echocardiography.
  Interventions: Device: transesophageal echocardiography (hTEE)
- OR-Cardiovascular: Requiring non-isolated cardiac surgery for repair of thoracic aortic aneurysm. Hemodynamic monitoring with transesophageal echo and hemodynamic support/ interventions include volume resuscitation, vasopressors, and positive inotropes. The Anesthesiologist may or may not use the information provided by the transesophageal echocardiography.
  Interventions: Device: transesophageal echocardiography (hTEE)

INTERVENTIONS:
Device: transesophageal echocardiography (hTEE) — Hemodynamic interventions include volume resuscitation, vasopressors and positive inotropes. Anesthesiologist may or may not use the information provided by the transesophageal echocardiography.
  Other Names: hTEE

SUMMARY:
The gold standard in hemodynamic evaluation has been the combined use of echocardiography and right heart catheterization. Fall backs to echocardiography are its time consumption and requirement for specialist interpretation while the Swan-Ganz® catheter shows a poor correlation of central venous pressure to volume status and provides indirect and difficult to interpret measurements in patients with unique pathophysiological states.

Next generation continuous hemodynamic transesophageal echocardiography (hTEE®) is being increasingly utilized to assist with complex resuscitations and to monitor the hemodynamic profiles of critically ill patients. hTEE is proving to be an essential diagnostic, therapeutic and monitoring tool for the rapid evaluation of the hemodynamic state in the critically ill patient and or hemodynamically compromised patient.

The purpose of this observational study is to evaluate the role of hTEE in clinical decision-making in 30 patients recruited from OR-Trauma and in 30 patients from the Cardiovascular-OR. Hemodynamic trans-esophageal echocardiography (hTEE) incorporates an FDA-approved miniaturized, disposable probe for continuous use in patients for up to 72 hours. This device has been used for postoperative assessment in the ICU for several years with successful placement of probes and without any adverse incidents.

The probe allows for the rapid, intermittent or continuous evaluation of bi-ventricular function, volume status and valve function at bedside or intraoperatively. It also allows for the evaluation of pericardial effusions and or the exclusion of pericardial tamponade.

DETAILED DESCRIPTION:
The device can evaluate trans-valvular flow as well as valvular regurgitation with the use of the color flow function. In many situations hTEE enables imaging not feasible by transthoracic echocardiography due to wounds, dressings, lines or edema.

The hTEE does not provide the visual acuity and detail of formal TEE, but it has the advantage of requiring a significantly smaller probe (hence the decreased risk of possible injury) with the ability of providing rapid, repeatable and sequential assessment by caregivers intraoperatively or at the bedside.

Data will be reviewed for outcome measures comparing efficiency, accuracy and clinical decision making capability of the FDA approved hTEE cardiac monitoring system vs. the standard of care Swan-Ganz/ echocardiographic information for publication. The ultimate goal will be to demonstrate whether or not after implementation of probes in surgical trauma and CVICU patients, there is a difference in:

1. Mortality and Morbidity
2. Organ dysfunction and failure
3. Blood product administration
4. Length of ICU stay
5. Hospital stay

2. Study Design and Statistical Procedures This is a two phase, single center, non-blinded, non-randomized, observational and retrospective study to be carried out at Memorial Hermann Hospital. The data from the hTEE study group will be compared to the control group (in-house OR-Trauma and CV surgery databases) and will be analyzed on a patient to patient basis for its impact on clinical decision-making.

Based upon our literature review, we hypothesize that hTEE will help guide point-of-care management upwards of 75 percent of cases. A decrease in iatrogenic complications from inappropriate blood product administration, volume resuscitation and or drug intervention based off of antiquated protocols and inaccurate technology is expected. Its use may benefit the hospital financially by decreasing the incidence of organ failure and mortality and allowing for the fulfillment of discharge criteria earlier from the hospital.

3. Study Procedures

1. Initiation A. Development of protocol and datasheet. (1 month) B. Training of anesthesia attendings, fellows, residents and technicians. (1 month) C. Formal presentation at Grand rounds. (1 month)
2. OR- Trauma/ CVICU:

   A. Training of the primary proceduralists. Board runners - 892 office. (1 month) B. Recording of real-time hemodynamic transesophageal echocardiographic movies of 60 patients. (3 months) C. Image analysis for clinical decision making with research assistants. (3 months)
3. Database retrospective review of above stated endpoints. (3 months)

   After admission to the OR and fulfillment of inclusion criteria, the hTEE probe will be placed by a trained attending or fellow as per standard care. A standardized exam will be performed that includes a: (1) superior vena cava view, (2) trans-esophageal four-chamber view and a (3) trans-gastric short axis view.

   As per current standard care, the information will be documented in the medical record and discussed with the PI, key study personnel and the patient's physician.

   For the purpose of the study, we will document carefully what impact the hTEE assessment has on the management plan on the first 60 patients who meet criteria and compare results to the standard of care use of CVP/ Echocardiography combination in terms of clinical decision making. Subsequent hTEE assessments will be made sequentially as clinically indicated, and the information obtained will be analyzed in the same way. All images will be stored for clinical interpretation on the machine itself, which is accessible to authorized personnel only. All patient data that is collected for the study will be coded; No subject identifiers will be recorded on study forms. See the privacy and confidentiality section for details.
4. Study Drugs or Devices: N/A
5. Study Instruments: N/A
6. Study Subjects:

Inclusion criteria:

• All study subjects 18 to 85 years old.

* OR-Trauma patients Presenting w/ hemodynamic instability. W/ expected intubation greater than 24 hours.
* CVICU patients Requiring non-isolated cardiac and vascular surgery

Exclusion criteria:

Current or previous esophageal injury

ELIGIBILITY:
Inclusion Criteria:

* • All study subjects 18 to 85 years old.

  * OR-Trauma patients Presenting w/ hemodynamic instability. W/ expected intubation greater than 24 hours.
  * CVICU patients (Cardiovascular Intensive Care Unit) Requiring non-isolated cardiac and vascular surgery

Exclusion Criteria:

* Current or previous esophageal injury

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients 18 to 85 years of age requiring hemodynamic monitoring during surgery for traumatic injury or non-isolated cardiac and vascular procedures.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Mortality and Morbidity | 30 days
  Comparing 30 day mortality and morbidity

SECONDARY OUTCOMES:
Organ dysfunction and failure | 30 days
  Comparing 30 day organ dysfunction and failure
Blood product administration | 48 hours
  Comparing Blood product administration during initial 48 hours
Length of ICU stay | 30 days
  Comparing Length of ICU stay
Hospital stay | 30 days
  Comparing Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Wegner, MD, Principal Investigator — The University of Texas Health Science Center, Houston

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vieillard-Baron A, Slama M, Mayo P, Charron C, Amiel JB, Esterez C, Leleu F, Repesse X, Vignon P. A pilot study on safety and clinical utility of a single-use 72-hour indwelling transesophageal echocardiography probe. Intensive Care Med. 2013 Apr;39(4):629-35. doi: 10.1007/s00134-012-2797-4. Epub 2013 Jan 4. PMID 23287876
- [Background] Gouveia V, Marcelino P, Reuter DA. The role of transesophageal echocardiography in the intraoperative period. Curr Cardiol Rev. 2011 Aug;7(3):184-96. doi: 10.2174/157340311798220511. PMID 22758616
- [Background] Treskatsch S, Balzer F, Knebel F, Habicher M, Braun JP, Kastrup M, Grubitzsch H, Wernecke KD, Spies C, Sander M. Feasibility and influence of hTEE monitoring on postoperative management in cardiac surgery patients. Int J Cardiovasc Imaging. 2015 Oct;31(7):1327-35. doi: 10.1007/s10554-015-0689-8. Epub 2015 Jun 6. PMID 26047772